CLINICAL TRIAL: NCT04560439
Title: METFIT Program - A Pilot Study Exploring the Feasibility of a Diabetes Prevention Program (DPP)-Based Lifestyle Modification Intervention to Reduce Insulin Resistance in Breast Cancer Survivors
Brief Title: Diabetes Prevention Program (METFIT) in Reducing Insulin Resistance in Stage I-III Breast Cancer Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19447; NCI-2020-04551 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19447 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-09-10; First posted 2020-09-23 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Early-Stage Breast Carcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (METFIT program) (Experimental): Patients undergo METFIT program for 16 sessions over 6 months.
  Interventions: Dietary Supplement: Dietary Intervention

INTERVENTIONS:
Dietary Supplement: Dietary Intervention — Undergo METFIT program
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions

SUMMARY:
This trial studies how well a diabetes prevention program (METFIT) works in reducing insulin resistance in stage I-III breast cancer survivors. METFIT program, a diet and lifestyle intervention, utilizes intermittent fasting to reduce insulin resistance in insulin resistant breast cancer survivors. Intermittent fasting has been shown to have benefits for patients undergoing cancer therapy by improving symptoms such as fatigue in breast cancer patients. Intermittent fasting has also shown potential for decreasing the risk of breast cancer coming back (recurrence). This trial is being done to determine if METFIT program can be successfully and effectively implemented to reduce insulin resistant in breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility of the METFIT Program - a 6-month modified Diabetes Prevention Program (DPP)-based lifestyle modification intervention that utilizes intermittent fasting (IF) aimed at reducing insulin resistance (IR) in insulin resistant breast cancer survivors.

SECONDARY OBJECTIVE:

I. To estimate an effect size of the effectiveness of the METFIT Program in reducing IR in insulin resistant breast cancer survivors.

OUTLINE:

Patients undergo METFIT program for 16 sessions over 6 months.

After completion of study treatment, patients are followed up for 40 days.

ELIGIBILITY:
Inclusion Criteria:

* Women who have been treated definitively for early stage breast cancer (I-III) and are 60-180 days from completion of chemotherapy, radiation and surgery regardless of hormonal status
* Demonstrated at least a 10% weight gain since being diagnosed with breast cancer
* Demonstrated IR by having a Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) score of >= 2.0
* Demonstrated IR manifested by meeting criteria for metabolic equivalent (MetS) as defined by modified criteria of the National Cholesterol Education Program Adult Treatment Panel (NCEP ATP III) (2005 version) and the World Health Organization (WHO) which includes:

  * Dysregulation of glucose homeostasis demonstrated by a glycosylated hemoglobin (HbA1c) >= 6.5%; OR fasting plasma glucose >= 126 mg/dl (7.0 mmol/L) OR random plasma glucose >= 200 mg/dL (11.1 mmol/L)
  * Plus two of any of the following:

    * Waist circumference in men >= 40 inches and in women >= 35 inches
    * Elevated triglycerides >= 150 mg/dL
    * Low high-density lipoprotein (HDL) cholesterol in men < 40 mg /dL and in women < 50 mg/dL or taking statin medication
    * Elevated blood pressure defined by a systolic pressure >= 130 of a diastolic pressure >= 85 mm Hg or taking anti-hypertensive medication
    * Elevated fasting glucose >= 110 mg/dL
* Non-smoker (last use 6 months prior to enrollment into the study)
* Documented informed consent of the participant and/or legally authorized representative
* Willingness to make substantial changes in their dietary and physical activity behavior
* Willingness to attend at 70% of the intervention sessions and 100% of the blood draws
* The effects of IF on the developing fetus of breast cancer survivors are unknown. For this reason, women of child bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating in the trial, should inform her treating physician immediately
* Willingness to weigh themselves weekly
* Willingness to wear a subcutaneous continuous glucose monitor
* Access to an electronic virtual teleconferencing device and capacity to utilize electronic teleconference technology

Exclusion Criteria:

* Use of any medication to treat diabetes mellitus
* Type 2 diabetes
* History of myocardial infarction or congestive heart failure within the previous 12 months prior to being screened for participation in the study
* Cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity
* Unstable cardiac disease as defined by one of the following:

  * Cardiac events such as myocardial infarction (MI) within the past 6 months
  * New York Heart Association (NYHA) heart failure class III-IV
  * Uncontrolled atrial fibrillation or hypertension
* History of vascular disease (e.g. deep vein thrombosis, stroke) within six months of starting the intervention
* Clinically significant uncontrolled illness
* Women who are pregnant or breastfeeding
* Any other condition (including psychosocial condition) that would, in the investigator's judgment, contraindicates the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Any other condition that would confound study results
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Fidelity | Up to week 8 of intervention
  The percentage of the cohort that has concordance of glucose trends with diet log to assess adherence to intermittent fasting regimen by week 8 of the intervention. Descriptive quantitative statistics will be used to report fidelity.
Retention | Up to 6 months
  Defined as the rate of participants that complete the intervention and post intervention assessments. Attendance percentage of blood draws and body measurements at both time points. Descriptive quantitative statistics will be used to report retention.

SECONDARY OUTCOMES:
Change in insulin resistance (IR) | Baseline to 6 months
  Assessed by Homeostatic Model Assessment of Insulin Resistance [HOMA-IR]). The HOMA-IR scores of each subject will be compared to their HOMA-IR scores after the intervention using a paired t-test analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Raynald Samoa, Principal Investigator — City of Hope Medical Center